CLINICAL TRIAL: NCT04718831
Title: Spirulina (FEM-102) Supplement to Chronic Hepatitis B Patients With High Levels of Quantitative Hepatitis B Surface Antigen
Brief Title: Spirulina (FEM-102) Supplement to Chronic Hepatitis B Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Far East Bio-Tec Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201810002
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis b
Keywords: Spirulina; Antigen
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (Other): Did not take nutritious food
  Interventions: Dietary Supplement: Spirulina
- General dose (Experimental): Taking 6g spirulina
  Interventions: Dietary Supplement: Spirulina
- Double dose (Experimental): Taking 12g spirulina
  Interventions: Dietary Supplement: Spirulina

INTERVENTIONS:
Dietary Supplement: Spirulina — Spirulina, as demonstrated in previous researches in vitro and in animals, can regulate immunity, enhance anti-virus activity, lower inflammation response and slower tumor progression. Liver function and liver fibrosis is improved by Spirulina as well. In our recent clinical trial, hepatitis B patients that received anti-virus medicine orally and was supplemented with Spirulina FEM-102 showed lower qHBsAg, reflecting the clearance of cccDNA. It might be related to immune modulation against HBV, which is induced by Spirulina.

SUMMARY:
Hepatocellular carcinoma (HCC), listed among lung and breast cancers as the top-ten cancer in 2016 Taiwan, is the second most prevalent cancer, just one place below colon cancer. Due to mass hepatitis B vaccination and the screening and therapeutic plan against hepatitis B and C viruses (HBV and HCV, respectively), the incidence of liver cancer drops significantly, however, still around twenty out of per hundred thousand population die from liver cancer each year. For patients suffering HBV and HCV, the prevention of HCC is a crucial health issue.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), listed among lung and breast cancers as the top-ten cancer in 2016 Taiwan, is the second most prevalent cancer, just one place below colon cancer. Due to mass hepatitis B vaccination and the screening and therapeutic plan against hepatitis B and C viruses (HBV and HCV, respectively), the incidence of liver cancer drops significantly, however, still around twenty out of per hundred thousand population die from liver cancer each year. For patients suffering HBV and HCV, the prevention of HCC is a crucial health issue.

The cause of HCC is mainly related to the hepatitis of HBV or HCV infection and subsequent cirrhosis. The population of HBV carrier is over 350 million in the world, three-fourths of them live in Asia-Pacific area. Therefore, hepatitis B may be the leading cause of HCC. For Taiwanese people born before 1986, the prevalence rate of hepatitis B is extremely high as 15-20%, and around 80% of HCC patients are also HBV carriers. In the past 20 years, for patients suffering with high level of HBV during immune clearance phase, immune residual inactive phase, reactivation phase and cirrhosis, our national health insurance cover the cost of interferon or other oral anti-virus medicine with defined criteria, dramatically lowering the risk of HCC developed from hepatitis B.

In previous clinical trial, some carriers showed high incidence of HCC when their quantitative hepatitis B surface antigen (qHBsAg) is high, especially when it is higher than 2000 IU/ml. The risk of HCC is still five-fold higher when the serum qHBsAg is above 1000 IU/ml. Therefore, it's important to explore novel intervention lowering qHBsAg.

Spirulina, as demonstrated in previous researches in vitro and in animals, can regulate immunity, enhance anti-virus activity, lower inflammation response and slower tumor progression. Liver function and liver fibrosis is improved by Spirulina as well. In our recent clinical trial, hepatitis B patients that received anti-virus medicine orally and was supplemented with Spirulina FEM-102 showed lower qHBsAg, reflecting the clearance of cccDNA. It might be related to immune modulation against HBV, which is induced by Spirulina.

Most chronic hepatitis patients do not meet most criteria of intervention according to our current guidelines. Since we already confirmed that Spirulina supplement can lower qHBsAg in treated patients, in this study we aim to understand whether Spirulina FEM-102, which regulate immunity against HBV as shown by the lowered qHBsAg, can lower the risk of HCC development of untreated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic hepatitis B do not take oral antiviral drugs.
2. Ages between 20 and 75.
3. High concentration of qHBsAg. qHBsAg≧1000 IU/ mL

Exclusion Criteria:

1. People allergic to seefood.
2. Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
HBV DNA | 6 months
  The change of HBV DNA during six months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shun Wu, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirahashi T, Matsumoto M, Hazeki K, Saeki Y, Ui M, Seya T. Activation of the human innate immune system by Spirulina: augmentation of interferon production and NK cytotoxicity by oral administration of hot water extract of Spirulina platensis. Int Immunopharmacol. 2002 Mar;2(4):423-34. doi: 10.1016/s1567-5769(01)00166-7. PMID 11962722
- [Background] Yakoot M, Salem A. Spirulina platensis versus silymarin in the treatment of chronic hepatitis C virus infection. A pilot randomized, comparative clinical trial. BMC Gastroenterol. 2012 Apr 12;12:32. doi: 10.1186/1471-230X-12-32. PMID 22497849
- [Background] Pham TX, Park YK, Bae M, Lee JY. The Potential Role of an Endotoxin Tolerance-Like Mechanism for the Anti-Inflammatory Effect of Spirulina platensis Organic Extract in Macrophages. J Med Food. 2017 Mar;20(3):201-210. doi: 10.1089/jmf.2016.0119. Epub 2017 Jan 25. PMID 28121488
- [Background] Munster VJ, Baas C, Lexmond P, Waldenstrom J, Wallensten A, Fransson T, Rimmelzwaan GF, Beyer WE, Schutten M, Olsen B, Osterhaus AD, Fouchier RA. Spatial, temporal, and species variation in prevalence of influenza A viruses in wild migratory birds. PLoS Pathog. 2007 May 11;3(5):e61. doi: 10.1371/journal.ppat.0030061. PMID 17500589